CLINICAL TRIAL: NCT06627608
Title: Treatment Prioritisation and Cost-Effectiveness Analysis for HBV Cure - Real-World Evidence from a Territory-Wide Cohort
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Grace Lai Hung Wong, Professor, Chinese University of Hong Kong
Other Study IDs: CEA for HBV cure
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Chronic Hepatitis B
Keywords: Cost-Effectiveness Analysis; HBV Cure
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
A number of hepatitis B virus (HBV) cure regimens including antisense oligonucleotide (ASO) and small interfering RNA (siRNA) are under vigorous clinical development and the efficacy and safety will soon be available for regulatory approval. Patients most in need should be prioritised to receive HBV cure regimen to maximise its clinical benefits and speed up hepatitis elimination.

DETAILED DESCRIPTION:
A territory-wide cohort study of all patients with chronic hepatitis B who have achieved functional cure of HBV. Real-world data will be used to estimate the risk of HCC, hepatic decompensation, and liver-related death for the subsequent simulation of HCC risk in particular populations of patients who achieved HBV cure. Literature search also be performed in parallel to cross-validate the estimates in untreated patients, and treated patients with incomplete or complete viral suppression with different stages of fibrosis based on existing literature. An optional systematic review and meta-analysis may be performed the address these issues.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic hepatitis B, i.e. hepatitis B surface antigen (HBsAg) or HBV DNA positive for two times at least 6 months apart, AND
2. Patients achieved HBV cure, i.e. HBsAg turned negative
3. Aged 18 years old or above.

Exclusion Criteria:

1. Patients with missing age and gender
2. Serious medical illnesses or malignancy with life expectancy <1 year
3. Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients with chronic hepatitis B, i.e. hepatitis B surface antigen (HBsAg) or HBV DNA positive for two times at least 6 months apart, AND
  2. Patients achieved HBV cure, i.e. HBsAg turned negative
  3. Aged 18 years old or above.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence rates of a composite endpoint of hepatic events, including hepatocellular carcinoma (HCC), cirrhotic complications and liver-related death | 20 years
  This would be the first step to get the estimated incidence rates of these clinical events to facilitate to subsequent modelling of the impact of different estimated rates of HBV cure on the overall incidence of liver outcomes.

SECONDARY OUTCOMES:
Economic burden | 20 years
  To determine the economic burden for managing HCC, hepatic event and liver-related death after an different possible increased rate of functional cure under new HBV cure regimens.
Partial HBV cure | 20 years
  To evaluate the impact of increased partial cure (sustained HBV DNA suppression without HBsAg loss after completing a finite course of antiviral treatment) on the incidence of HCC, hepatic event and liver-related death after an different possible reduction of HBsAg levels under new HBV cure regimens.
Establish the most desirable cost range | 20 years
  To establish the most desirable cost range for the first approved HBV cure regimen using Hong Kong and the Greater Bay Area (GBA) as the examples (with the healthcare cost variations in different regions of GBA taken into account).
Healthcare resources saving | 20 years
  To determine the healthcare resources saving from the reduced incidence of HCC, hepatic event and liver-related death after an different possible increased rate of functional cure under new HBV cure regimens.

IPD SHARING:
Plan to Share IPD: No